CLINICAL TRIAL: NCT01867489
Title: A Qualitative Study Into How Patients With Cancer Deal With Chemotherapy-Related Side Effects at Home
Brief Title: A Qualitative Study Into How Patients Deal With Chemotherapy-related Side Effects at Home
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Annemarie Coolbrandt, Clinical Nurse Specialist Oncology, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: B322201214929
Record Dates: First submitted 2013-05-19; First posted 2013-06-04 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Exploration of How Patients Deal With Side Effects From Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemotherapy, Cancer: Adult cancer patients (with any type of cancer) being treated with chemotherapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This qualitative study explores how patients deal with the side effects from chemotherapy at their home, what factors and ideas influence their symptom self-management and how professional caregivers contribute to the management of their symptoms at home. Data are collected through semi-structured interviews with adult patients treated with chemotherapy and analysed using a Grounded Theory approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients with (any type and any stage of) cancer who were undergoing chemotherapy treatment in an ambulatory setting or during short hospital stays
* Dutch speaking
* Able to provide informed consent and to participate in an interview

Exclusion Criteria:

* Patients who were in the first 2 cycles of treatment
* Patients for whom an interview was considered physically, mentally and/or emotionally too burdensome.
* Patients who had reported not to experience any side effect from treatment at all

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
patient's experience | one interview during the course of treatment, i.e. one timepoint between 2 months after the start of chemotherapy and the end of the patient's treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium